CLINICAL TRIAL: NCT05566639
Title: A Phase 3, Randomized, Observer-blind, Active-controlled Study to Evaluate the Safety and Efficacy of mRNA-1010 Candidate Seasonal Influenza Vaccine in Adults 50 Years and Older
Brief Title: A Study of mRNA-1010 Seasonal Influenza Vaccine in Adults 50 Years Old and Older
Status: Completed | Phase: Phase 3 | Type: Interventional
Sponsor: ModernaTX, Inc. (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Triple | Purpose: Prevention
Other Study IDs: mRNA-1010-P302; 2022-001638-12 (EudraCT Number)
Record Dates: First submitted 2022-09-30; First posted 2022-10-04 (Actual); Results first posted 2025-01-16 (Actual); Last update posted 2025-01-16 (Actual); Status verified 2024-12

CONDITIONS: Seasonal Influenza
Keywords: Flu; Influenza; Vaccine; mRNA vaccine; mRNA-1010; Moderna
MeSH Terms: conditions — Influenza, Human | interventions — mRNA-1010 influenza vaccine

STUDY DESIGN:
Who Masked: Participant, Investigator, Outcomes Assessor
Oversight: FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (2):
- mRNA-1010 (Experimental): Participants will receive a single dose of mRNA-1010 by intramuscular (IM) injection on Day 1.
  Interventions: Biological: mRNA-1010
- Fluarix Quadrivalent (Active Comparator): Participants will receive a single dose of Fluarix Quadrivalent by IM injection on Day 1.
  Interventions: Biological: Fluarix Quadrivalent

INTERVENTIONS:
Biological: mRNA-1010 — Sterile liquid for injection
  Other Names: Seasonal influenza vaccine
  Arms: mRNA-1010
Biological: Fluarix Quadrivalent — Sterile suspension for injection.
  Other Names: Licensed quadrivalent inactivated seasonal influenza vaccine
  Arms: Fluarix Quadrivalent

SUMMARY:
The purpose of this study is to evaluate the safety and efficacy of mRNA-1010 in preventing seasonal influenza in adults 50 years and older.

ELIGIBILITY:
Inclusion Criteria:

* Investigator has assessed that the participant understands and is willing and physically able to comply with protocol mandated follow-up, including all procedures.

  * For female participants of childbearing potential: negative pregnancy test, adequate contraception or has abstained from all activities that could result in pregnancy for at least 28 days prior to the first dose on Day 1, and agreement to continue adequate contraception through 90 days following vaccine administration.

Exclusion Criteria:

* Participant has had close contact with someone with laboratory-confirmed influenza infection or with someone who has been treated with antiviral therapies for influenza (for example, Tamiflu®) within the past 5 days prior to the Screening visit.
* Participant has had close contact to someone with severe acute respiratory syndrome coronavirus 2 (SARS-CoV-2) infection or COVID-19 as defined by the US CDC or has had a positive SARS-CoV-2 test in the past 10 days prior to the Screening visit.
* Participant is acutely ill or febrile (temperature ≥38.0℃elcius [100.4°Fahrenheit]) 72 hours prior to or at the Screening visit or Day 1. Participants meeting this criterion may be rescheduled within the 28-day screening window.
* Participant has a history of a diagnosis or condition that, in the judgment of the investigator, is clinically unstable or may affect participant safety, assessment of safety endpoints, assessment of immune response, or adherence to study procedures.
* Reported history of congenital or acquired immunodeficiency, immunocompromising/ immunosuppressive condition, asplenia, or recurrent severe infections.
* Reported history of anaphylaxis or severe hypersensitivity reaction after receipt of any mRNA or influenza vaccines or any components of the mRNA or influenza vaccines, including egg protein.
* Participant has received systemic immunosuppressant drugs for >14 days in total within 180 days prior to the Screening visit (for glucocorticosteroids, ≥10 milligrams (mg)/day of prednisone or equivalent) or is anticipating the need for systemic immunosuppressive treatment at any time during participation in the study. Inhaled, nasal, and topical steroids are allowed.
* Participant has received any vaccine authorized or approved by local health agency ≤28 days prior to study intervention (Day 1) or plans to receive a vaccine authorized or approved by local health agency within 28 days before or after the study intervention.
* Participant is unaware whether they have received an influenza vaccine in the previous influenza season.
* Participant received a seasonal influenza vaccine or any other investigational influenza vaccine within 180 days prior to Day 1
* Participant has tested positive for influenza by local health authority-approved testing methods within 180 days prior to Day 1.
* Participant has donated ≥450 milliliters (mL) of blood products within 28 days prior to the Screening visit or plans to donate blood products during the study.

Note: Other inclusion and exclusion criteria may apply.

Min Age: 50 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 22502 (Actual)
Dates: Start 2022-09-14 (Actual); Primary Completion 2024-01-05 (Actual); Study Completion 2024-01-05 (Actual)

CONTACTS AND LOCATIONS:
Locations (231):
- United States (133):
  - North Alabama Research Center, LLC, Athens, Alabama
  - Lenzmeier Family Medicine, Glendale, Arizona
  - CCT Research, Phoenix, Arizona
  - Fiel Family and Sports Medicine/CCT Research, Tempe, Arizona
  - Noble Clinical Research, Tucson, Arizona
  - Lynn Institute of the Ozarks, Little Rock, Arkansas
  - Baptist Health Center for Clinical Research, Little Rock, Arkansas
  - Velocity Clinical Research, Banning, Banning, California
  - Hope Clinical Research, LLC, Canoga Park, California
  - Marvel Clinical Research, Huntington Beach, California
  - Velocity Clinical Research, Chula Vista, La Mesa, California
  - Velocity Clinical Research, San Diego, La Mesa, California
  - Velocity Clinical Research - Westlake, Los Angeles, California
  - Empire Clinical Research, Pomona, California
  - Artemis Institute for Clinical Research, Riverside, California
  - Benchmark Research-Texas, Riverside, California
  - Peninsula Research Associates (PRA), Rolling Hills Estates, California
  - Artemis Institute for Clinical Research, San Diego, California
  - Women's Health Care Research Corp., San Diego, California
  - Acclaim Clinical Research, San Diego, California
  - Medical Center for Clinical Research, San Diego, California
  - Shawn K Hassler MD, San Francisco, California
  - West Coast Research LLC, San Ramon, California
  - Velocity Clinical Research, Denver, Denver, Colorado
  - Arthritis & Rheumatology - Clinic of Northern Colorado, Fort Collins, Colorado
  - Longmont Medical Research Network, Longmont, Colorado
  - Nature Coast Clinical Research, LLC - Crystal River, Crystal River, Florida
  - Floridian Clinical Research, Hialeah, Florida
  - Homestead Associates in Research,Inc, Hialeah, Florida
  - Broward Research Group, Hollywood, Florida
  - Citrus Cardiology Consultants, Inverness, Florida
  - Encore Research Group-Jacksonville Center for Clinical Resea, Jacksonville, Florida
  - Health Awareness, Inc, Jupiter, Florida
  - Multi-Therapeutic Research Associates, Inc., Lake City, Florida
  - Accel Research Sites - Lakeland, Lakeland, Florida
  - ARS - Meridien Research, Maitland, Florida
  - South Florida Research Center, Inc., Miami, Florida
  - Suncoast Research Associates Trials, LLC, Miami, Florida
  - Miami centre of clinical research, Miami, Florida
  - Clinical Trials of Florida, LLC, Miami, Florida
  - Global Health Research Center, Miami Lakes, Florida
  - Innovation Medical Research Center,inc, Palmetto Bay, Florida
  - New Tampa Health, Inc, Tampa, Florida
  - Tekton Research, Inc., Chamblee, Georgia
  - Southeast Regional Research Group, Columbus, Georgia
  - iResearch Atlanta, LLC, Decatur, Georgia
  - In-Quest Medical Research, Norcross, Georgia
  - Mount Vernon Clinical Research, Sandy Springs, Georgia
  - Meridian Clinical Research - Savannah, Savannah, Georgia
  - Clinical Research Atlanta, Stockbridge, Georgia
  - Velocity Clinical Research - Boise, Meridian, Idaho
  - Great Lakes Clinical Trials LLC, Chicago, Illinois
  - Great Lakes Clinical Trials LLC, Gurnee, Illinois
  - Chicago Health Medical Group, River Forest, Illinois
  - Velocity Clinical Research - Valparaiso, Valparaiso, Indiana
  - Meridian Clinical Research - Dakota Dunes, Sioux City, Iowa
  - Johnson County Clin-Trials (JCCT), Lenexa, Kansas
  - Heartland Research Associates LLC, Newton, Kansas
  - Alliance for Multispecialty Research, Wichita, Kansas
  - Meridian Clinical Research, Baton Rouge, Louisiana
  - MedPharmics, Covington, Louisiana
  - Medpharmics, LLC, Metairie, Louisiana
  - Nathan H Fischman MD LLC, New Orleans, Louisiana
  - Privia Medical Group, Annapolis, Maryland
  - Rockville Internal Medicine Group, Rockville, Maryland
  - Delricht Research, Springfield, Massachusetts
  - DM Clinical Research - Detroit, Southfield, Michigan
  - Paul G Matherne MD, Biloxi, Mississippi
  - DELRICHT RESEARCH at GULFPORT MEMORIAL, Gulfport, Mississippi
  - National Medical University and Embryonic Tissues Center EmC, Springfield, Missouri
  - Sundance Clinical Research, LLC, St Louis, Missouri
  - Montana Medical Research, Inc, Missoula, Montana
  - CCT Research at Skyline Medical Center, PC, Elkhorn, Nebraska
  - CCT Research / Methodist Physicians Clinic, Prairie Fields Family Medicine, PC, Fremont, Nebraska
  - Meridian Clinical Research, Grand Island, Nebraska
  - Be Well Clinical Studies, LLC, Lincoln, Nebraska
  - Medpace, Inc. - Clinical Pharmacology Unit (CPU), Norfolk, Nebraska
  - Meridian Clinical Research, Norfolk, Nebraska
  - Papillon Research Centre, Omaha, Nebraska
  - Meridian Clinical Research - Omaha, Omaha, Nebraska
  - Midwest Regional Health Services, LLC/CCT Research, Omaha, Nebraska
  - CCT Research, Las Vegas, Nevada
  - Clinical Research Center of Nevada LLC, Las Vegas, Nevada
  - Santa Rosa Medical Centers of Nevada/ CCT Research, Las Vegas, Nevada
  - Las Vegas Clinical Trials, LLC, North Las Vegas, Nevada
  - United Medical Associates, Binghamton, New York
  - Rochester Clinical Research, Inc, Rochester, New York
  - Velocity Clinical Research - Syracuse, Syracuse, New York
  - Tryon Medical Group, Charlotte, North Carolina
  - Carolina Institute for Clinical Research, Fayetteville, North Carolina
  - Diabetes & Endocrinology Consultants, Morehead City, North Carolina
  - M3 Wake Research, Inc., Raleigh, North Carolina
  - PMG Research of Wilmington, Wilmington, North Carolina
  - Trial Management Associates, Wilmington, North Carolina
  - Wake Forest Baptist Medical Center, Winston-Salem, North Carolina
  - Radiant Research, Akron, Ohio
  - Sterling Research Group, Cincinnati, Ohio
  - CTI Clinical Research Center, Cincinnati, Ohio
  - Velocity Clinical Research - Cincinnati, Cincinnati, Ohio
  - Lynn Health Science Institute, Oklahoma City, Oklahoma
  - Delricht Research Tulsa, Tulsa, Oklahoma
  - Platinum Research Network, LLC, Yukon, Oklahoma
  - Velocity Clinical Research - Grants Pass, Grants Pass, Oregon
  - Velocity Clinical Resarch - Medford, Medford, Oregon
  - Velocity Clinical Research - Providence, Warwick, Rhode Island
  - Velocity Clinical Research, Greenville, Anderson, South Carolina
  - Velocity Clinical Research - Columbia, Columbia, South Carolina
  - Velocity Clinical Research, Gaffney, Gaffney, South Carolina
  - Velocity Clinical Research - Greenville, Greenville, South Carolina
  - Carolina Health Specialists, Myrtle Beach, South Carolina
  - Spartanburg Regional Health Services, Spartanburg, South Carolina
  - Black Hills Center for American Indian Health, Rapid City, South Dakota
  - Delricht Research, Hendersonville, Tennessee
  - Tekton Research, Inc, Austin, Texas
  - Platinum Research Network, LLC, Beaumont, Texas
  - Zenos Clinical Research, Dallas, Texas
  - Benchmark Research, Fort Worth, Texas
  - DM Clinical Research, Houston, Texas
  - Texas Center for Drug Development, Inc., Houston, Texas
  - DELRICHT RESEARCH at ZOMNIR FAMILY MEDICINE, McKinney, Texas
  - Research Your Health, Plano, Texas
  - Epic Medical Research, LLC, Red Oak, Texas
  - Clinical Trials of Texas, Inc, San Antonio, Texas
  - DM Clinical Research, Sugar Land, Texas
  - Breco Research - A Tarheel Clinical Research Site, Sugar Land, Texas
  - Cope Family Medicine, Bountiful, Utah
  - Olympus Family Medicine/CCT Research, Holladay, Utah
  - CenExel - JBR, Salt Lake City, Utah
  - South Ogden Family Medicine clinic/CCT, South Ogden, Utah
  - Velocity Clinical Research - Salt Lake City, West Jordan, Utah
  - Meridian Clinical Research, Portsmouth, Virginia
  - Clinical Research Partners, LLC, Richmond, Virginia
  - Lakeview Medical Center, Suffolk, Virginia
- Bulgaria (6):
  - MHAT Sveti Ivan Rilski, Kozloduy
  - MC City Clinic Sveti Georgi - Montana, Montana
  - MHAT "Dr. Stamen Iliev, Montana
  - Medical Center Medconsult Pleven, Pleven
  - Military Medical Academy, Sofia
  - SHAT of Pneumo-phthisiatric diseases - Sofia District, Sofia
- Canada (24):
  - Aggarwal and Associates LTD, Brampton
  - Aviva Clinical Trials Group Inc, Burlington
  - Hamilton Medical Research Group, Hamilton
  - Okanagan Clinical Trials, Kelowna
  - Centricity Research Quebec City, Lévis
  - Milestone Research Inc., London
  - Yang Medicine, Ottawa
  - LMC Manna, Pointe-Claire
  - DIEX Research Quebec Inc., Québec
  - Alpha Recherche Clinique Inc, Québec
  - Clinique de Lebourgneuf, Québec
  - Clinique spécialisée en allergie - Allergy/Immunology/Asthma/Mpoc, Québec
  - Diex Research Sherbrooke Inc, Québec
  - Central Alberta Research Clinic, Red Deer
  - Diex Recherche - Joilette - HyperCore - PPDS, Saint-Charles-Borromée
  - Glencar Medical Inc., Sarnia
  - Canadian Phase Onward Inc., Toronto
  - LMC, Toronto
  - Manna Research, Toronto
  - Medicine Professional Corporation, Toronto
  - Toronto Western Hospital, Toronto
  - Diex Recherche Trois-Rivières, Trois-Rivières
  - Colchester East Hants Health Authority - Colchester Regional, Truro
  - Diex Recherche Victoriaville, Victoriaville
- Denmark (3):
  - Aarhus Universitetshospital, Århus N
  - Odense University Hospital, Odense
  - Sjællands UniHosp, Roskilde - Medicine and Infectious Diseases, Roskilde
- Estonia (4):
  - Center for Clinical and Basic Research, Tallinn
  - Innomedica OÜ, Tallinn
  - Merelahe Family Doctors Centre, Tallinn
  - Clinical Research Center, Tartu
- Germany (22):
  - Berliner Centrum für Reise- und Tropenmedizin, Berlin
  - Emovis GmbH, Berlin
  - Klinische Forschung Berlin-Mitte GmbH, Berlin
  - Klinische Forschung Berlin, Berlin
  - University Hospital Cologne AöR, Cologne
  - Klinische Forschung Dresden GmbH, Dresden
  - Medizentrum Essen Borbeck, Essen
  - IKF Pneumologie, Frankfurt
  - Infektiologikum Frankfurt-Sachsenhausen, Frankfurt
  - Studienzentrum Dr. Keller, Frankfurt am Main
  - Clinical Research Hamburg GmbH, Hamburg
  - Klinische Forschung Hamburg GmbH, Hamburg
  - Klinische Forschung Hannover-Mitte GmbH, Hanover
  - Siteworks GmbH, Hanover
  - Siteworks GmbH, Heidelberg
  - Synexus Clinical Research GmbH, Leipzig
  - Praxis Illies, Magdeburg
  - Dermatologie Quist, Mainz
  - Praxis Schaum, Oldenburg
  - Klinische Forschung Schwerin GmbH, Schwerin
  - Hautarztpraxis Leitz & Kollegen, Stuttgart
  - Studienzentrum Brinkum, Wardenburg
- Netherlands (2):
  - Leids Universitair Medisch Centrum (LUMC), Leiden
  - Universitair Medisch Centrum (UMC) Utrecht - Julius Center for Health Sciences and Primary Care, Utrecht
- Poland (12):
  - Centrum Medyczne Pratia Bydgoszcz, Bydgoszcz
  - Centrum Medyczne Plejady, Krakow
  - Krakowskie Centrum Medyczne Sp. z o.o., Krakow
  - Centrum Medyczne AMED Oddzial w Lodzi, Lodz
  - ETG Lublin, Lublin
  - KO-MED Centra Kliniczne Lublin II, Lublin
  - ETG Skierniewice, Skierniewice
  - Centrum Innowacyjnych Terapii Sp. z o.o., Warsaw
  - Provita Centrum Medyczne Sp. z o.o., Warsaw
  - RCMed, Warsaw
  - ETG Zamosc, Zamość
  - KO-MED Centra Kliniczne Sp. z o.o., Zamość
- Spain (6):
  - Hospital de Antequera, Antequera
  - Hospital Clinic De Barcelona, Barcelona
  - Hospital Santa Creu i Sant Pau - Research institut, Barcelona
  - Universitat Autonoma de Barcelona (UAB) - Institut d'Investigacio en Atencio Primaria Jordi Gol (IDIAP Jordi Gol), Barcelona
  - Hospital Alvaro Cunqueiro, Vigo
  - Hospital Povisa, Vigo
- Taiwan (7):
  - Kaohsiung Veterans General Hospital, Kaohsiung City
  - China Medical University Hospital - division of Rheumatology - Taichung, Taichung
  - National Cheng Kung University hospital, Tainan
  - National Taiwan University Hospital - Family Medicine, Taipei
  - Taipei Medical University - Taipei Medical University Hospital, Taipei
  - Taipei Medical University - WanFang Hospital, Taipei
  - Tri-Service General Hospital - Neihu Branch - Infectious Diseases, Taipei
- United Kingdom (12):
  - Royal United Hospital, Bath
  - Layton Medical Centre, Blackpool
  - Hull University Teaching Hospitals NHS Foundation trust, Hull
  - University Hospitals of Leicester-Leicester Royal Hospital, Leicester
  - Liverpool University Hospitals NHS Foundation Trust - Aintree University Hospital (Fazakerley Hospital), Liverpool
  - GST NHS Found, London
  - Newcastle University - Institute of Cellular Medicine (ICM), Newcastle
  - Panthera Biopartners - Manchester - multispeciality, Rochdale
  - Panthera Biopartners - Sheffield - multispeciality, Rochdale
  - Panthera Biopartners - Preston - multispeciality, Salford
  - Southampton General Hospital, Southampton
  - Royal Cornwall Hospitals Trust - Respiratory, Truro

RESULTS

PARTICIPANT FLOW:
Pre-assignment Details: A total of 22502 participants were randomized in this study, including 11252 participants in the mRNA-1010 group and 11250 participants in the Fluarix Quadrivalent group.
Groups:
- Fluarix Quadrivalent: Participants received a single dose of Fluarix Quadrivalent by intramuscular (IM) injection on Day 1.
- mRNA-1010: Participants received a single dose of mRNA-1010 by IM injection on Day 1.
Period: Overall Study
Arm/Group | Fluarix Quadrivalent | mRNA-1010
Started | 11250 | 11252
Full Analysis Set (All randomized participants who received any study intervention.) | 11199 | 11211
Safety Set (All randomized participants who received any study intervention. Participants were included in the vaccination group corresponding to the study intervention that they actually received.) | 11200 | 11210
Solicited Safety Set (All randomized participants who received any study intervention and contributed to any solicited AR data.) | 11160 | 11168
Per-Protocol (PP) Set (All participants in the Modified Intent-to-Treat (mITT) Set (all randomized participants who received any study intervention except those who discontinued from the study prior to 14 days following administration of study intervention) who did not have major protocol deviations that could adversely impact efficacy, for example, disease or therapeutic intervention that might cause suboptimal response to the study intervention.) | 11026 | 11055
PP Immunogenicity Set (PPIS) (All randomized participants in the biomarker subset who received any study intervention; had baseline and Day 29 antibody assessment via HAI assay; complied with the immunogenicity testing schedule, and had no major protocol deviations that impacted the immunogenicity assessment.) | 408 | 444
Completed | 10359 | 10359
Not Completed | 891 | 893
Not completed — Adverse Event | 1 | 1
Not completed — Serious Adverse Event | 1 | 3
Not completed — Death | 44 | 45
Not completed — Lost to Follow-up | 467 | 461
Not completed — Physician Decision | 45 | 44
Not completed — Protocol Deviation | 4 | 4
Not completed — Withdrawal by Subject | 277 | 271
Not completed — Other Than Specified | 52 | 64

BASELINE CHARACTERISTICS:
Population: Randomization Set included all participants who were randomized, regardless of the participant's treatment status in the study.
Groups:
- Fluarix Quadrivalent: Participants received a single dose of Fluarix Quadrivalent by IM injection on Day 1.
- Total: Total of all reporting groups
Arm/Group | Fluarix Quadrivalent | mRNA-1010 | Total
Number analyzed (Participants) | 11250 | 11252 | 22502
Age, Continuous [Mean (Standard Deviation); unit: years] | 63.8 (8.41) | 63.9 (8.36) | 63.9 (8.39)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 6281 | 6256 | 12537
  Male | 4969 | 4996 | 9965
Ethnicity (NIH/OMB) [Count of Participants; unit: Participants]
  Hispanic or Latino | 1837 | 1859 | 3696
  Not Hispanic or Latino | 9289 | 9273 | 18562
  Unknown or Not Reported | 124 | 120 | 244
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 55 | 57 | 112
  Asian | 280 | 254 | 534
  Native Hawaiian or Other Pacific Islander | 15 | 11 | 26
  Black or African American | 1986 | 1950 | 3936
  White | 8790 | 8850 | 17640
  More than one race | 37 | 48 | 85
  Unknown or Not Reported | 87 | 82 | 169

OUTCOME MEASURES:

1. Primary Outcome: Number of Participants With Solicited Local and Systemic Reactogenicity Adverse Reactions (ARs)
Description: Solicited ARs (local and systemic) were collected in an electronic diary (eDiary). Local ARs included: injection site pain, injection site erythema (redness), injection site swelling/induration (hardness), and axillary (underarm) swelling or tenderness ipsilateral to the side of injection. Systemic ARs included: fever, headache, fatigue, myalgia, arthralgia, nausea/vomiting, and chills. All solicited ARs considered causally related to injection were graded 0-4 (per Toxicity Grading Scale for Healthy Adult and Adolescent Volunteers Enrolled in Preventive Vaccine Clinical Trials); lower score indicates lower severity, and a higher score indicates greater severity. Note, not all solicited ARs were considered adverse events (AEs). The Investigator reviewed whether the solicited AR was also to be recorded as an AE. A Summary of serious AEs (SAEs) and nonserious AEs ("Other"), regardless of causality, is located in the "Reported Adverse Events" section.
Time Frame: 7 days post-vaccination
Population: Solicited Safety Set included all randomized participants who received any study intervention and contributed to any solicited AR data.
Measure: Count of Participants; unit: Participants
Arm/Group | Fluarix Quadrivalent | mRNA-1010
Number analyzed (Participants) | 11160 | 11168
Participants
  Any | 5620 | 7989
  Grade 1 | 3840 | 4433
  Grade 2 | 1535 | 3050
  Grade 3 | 245 | 500
  Grade 4 | 0 | 6

2. Primary Outcome: Number of Participants With Unsolicited Adverse Events (AEs)
Description: An unsolicited AE was an AE that was not solicited using a participant diary and that was communicated by a participant who has signed the informed consent. An AE was defined as any untoward medical occurrence associated with the use of a drug in humans, whether or not considered drug related. Any abnormal laboratory test result (hematology, clinical chemistry, or prothrombin time [PT]/partial thromboplastin time [PTT]) or other safety assessment (for example, electrocardiogram, radiological scan, vital sign measurement), including one that worsened from baseline and was considered clinically significant in the medical and scientific judgment of the Investigator was recorded as an AE. Number of participants with unsolicited AEs (SAEs and non-serious AEs) up to 28 days post-vaccination are reported in this outcome measure.
Time Frame: Up to 28 days post-vaccination
Population: Safety Set included all randomized participants who received any study intervention. Participants were included in the vaccination group corresponding to the study intervention that they actually received.
Measure: Count of Participants; unit: Participants
Arm/Group | Fluarix Quadrivalent | mRNA-1010
Number analyzed (Participants) | 11200 | 11210
Participants | 1495 | 1351

3. Primary Outcome: Number of Participants With Serious Adverse Events (SAEs), AEs of Special Interest (AESIs), Medically Attended AEs (MAAEs), and AEs Leading to Discontinuation
Description: An SAE was defined as any AE that resulted in death, was life-threatening, required inpatient hospitalization or prolongation of existing hospitalization, resulted in disability/permanent damage, was a congenital anomaly/birth defect, or was an important medical event. AESIs included thrombocytopenia, new onset of or worsening of the protocol specified neurologic diseases, anaphylaxis, and myocarditis/pericarditis. An MAAE is an AE that lead to an unscheduled visit to an healthcare practitioner. This included visits to a study site for unscheduled assessments (for example, abnormal laboratory follow-up, and/or coronavirus disease 2019 [COVID-19] and visits to healthcare practitioners external to the study site (for example, urgent care, primary care physician). Number of participants with SAEs, AESIs, MAAEs, and AEs leading to discontinuation up to the end of study (Day 361) are reported in this outcome measure.
Time Frame: Day 1 through Day 361 (Month 12)
Population: as for outcome 2
Measure: Count of Participants; unit: Participants
Arm/Group | Fluarix Quadrivalent | mRNA-1010
Number analyzed (Participants) | 11200 | 11210
Participants
  SAEs | 495 | 518
  AESIs | 13 | 10
  MAAEs | 3166 | 3126
  AEs Leading to Discontinuation | 47 | 49

4. Primary Outcome: Number of Participants With First Episode of RT-PCR-Confirmed Protocol-Defined Influenza-Like Illness (ILI) Caused by Any Seasonal Influenza A or B Virus Strains Regardless of Antigenic Match to Strains Selected for the Seasonal Vaccine
Description: Protocol-defined ILI: The presence of body temperature ≥37.5 degrees celsius (°C) (≥99.5 degrees fahrenheit [°F]), accompanied by at least one of the respiratory illness symptoms (sore throat, cough, sputum production, wheezing, or difficulty breathing) and a positive Reverse Transcription Polymerase Chain Reaction (RT-PCR) for influenza.
Time Frame: 14 days post-vaccination through Day 181 (Month 6)
Population: Per-Protocol (PP) Set included all participants in the Modified Intent-to-Treat (mITT) Set (all randomized participants who received any study intervention except those who discontinued from the study prior to 14 days following administration of study intervention) who did not have major protocol deviations that could adversely impact efficacy, for example, disease or therapeutic intervention that might cause suboptimal response to the study intervention.
Measure: Count of Participants; unit: Participants
Arm/Group | Fluarix Quadrivalent | mRNA-1010
Number analyzed (Participants) | 11026 | 11055
Participants | 142 | 140
Statistical Analysis 1: Comparison: Fluarix Quadrivalent vs mRNA-1010; Test type: Non-Inferiority — Noninferiority margin = 10%; p = 0.1715, Stratified Cox proportional hazards; Relative vaccine efficacy (rVE) = 1.7, 95% CI 2-sided [-24.1 to 22.2] — rVE = 100 * (1 - HR) % was defined as the percent reduction in the hazard (mRNA-1010 vs active comparator), where HR was the hazard ratio between mRNA-1010 vs the active comparator

5. Secondary Outcome: Number of Participants With First Episode of RT-PCR-Confirmed Protocol-Defined ILI Caused by Influenza A or B Strains With Similarity to Those Selected for the Seasonal Vaccine
Description: Protocol-defined ILI: The presence of body temperature ≥37.5°C (≥99.5°F), accompanied by at least one of the respiratory illness symptoms (sore throat, cough, sputum production, wheezing, or difficulty breathing) and a positive RT-PCR for influenza.
Time Frame: 14 days post-vaccination through Day 181 (Month 6)
Population: As pre-specified, the data for this outcome measure was not collected and analyzed.
Arm/Group | Fluarix Quadrivalent | mRNA-1010
Number analyzed (Participants) | 0 | 0

6. Secondary Outcome: Number of Participants With First Episode of RT-PCR-Confirmed Protocol-Defined ILI Caused by Influenza A or B Strains Antigenically Matched to the Vaccine Strains Selected for the Seasonal Vaccine
Description: as for outcome 5
Time Frame: 14 days post-vaccination through Day 181 (Month 6)
Population: PP Set included all participants in the mITT Set (all randomized participants who received any study intervention except those who discontinued from the study prior to 14 days following administration of study intervention) who did not have major protocol deviations that could adversely impact efficacy, for example, disease or therapeutic intervention that might cause suboptimal response to the study intervention.
Measure: Count of Participants; unit: Participants
Arm/Group | Fluarix Quadrivalent | mRNA-1010
Number analyzed (Participants) | 11026 | 11055
Participants | 85 | 75

7. Secondary Outcome: Number of Participants With First Episode of RT-PCR Confirmed United States (US) Centers for Disease Control and Prevention (CDC)-Defined ILI Caused by Any Influenza A or B Strains
Description: CDC-defined ILI: The presence of temperature ≥37.8°C [≥100°F], accompanied by at least one of the respiratory illness symptoms (cough and/or sore throat) and a positive RT-PCR for influenza.
Time Frame: 14 days post-vaccination through Day 181 (Month 6)
Population: as for outcome 6
Measure: Count of Participants; unit: Participants
Arm/Group | Fluarix Quadrivalent | mRNA-1010
Number analyzed (Participants) | 11026 | 11055
Participants | 70 | 70

8. Secondary Outcome: Number of Participants With First Episode of RT-PCR CDC-Defined ILI Caused by Influenza A or B Strains With Similarity to Vaccine Strains
Description: as for outcome 7
Time Frame: 14 days post-vaccination through Day 181 (Month 6)
Population: As pre-specified, the data for this outcome measure was not collected and analyzed.
Arm/Group | Fluarix Quadrivalent | mRNA-1010
Number analyzed (Participants) | 0 | 0

9. Secondary Outcome: Number of Participants With First Episode of RT-PCR CDC-Defined ILI Caused by Influenza A or B Strains That Were Antigenically Matched to Vaccine Strains
Description: as for outcome 7
Time Frame: 14 days post-vaccination through Day 181 (Month 6)
Population: as for outcome 6
Measure: Count of Participants; unit: Participants
Arm/Group | Fluarix Quadrivalent | mRNA-1010
Number analyzed (Participants) | 11026 | 11055
Participants | 44 | 38

10. Secondary Outcome: Number of Participants With First Episode of Culture-Confirmed Protocol-Defined ILI Caused by Any Seasonal Influenza A or B Virus Strains Regardless of Antigenic Match to Strains Selected for the Seasonal Vaccine
Description: as for outcome 5
Time Frame: 14 days post-vaccination through Day 181 (Month 6)
Population: as for outcome 6
Measure: Count of Participants; unit: Participants
Arm/Group | Fluarix Quadrivalent | mRNA-1010
Number analyzed (Participants) | 11026 | 11055
Participants | 91 | 81

11. Secondary Outcome: Number of Participants With First Episode of Culture-Confirmed CDC-Defined ILI Caused by Any Seasonal Influenza A or B Virus Strains Regardless of Antigenic Match to Strains Selected for the Seasonal Vaccine
Description: as for outcome 7
Time Frame: 14 days post-vaccination through Day 181 (Month 6)
Population: as for outcome 6
Measure: Count of Participants; unit: Participants
Arm/Group | Fluarix Quadrivalent | mRNA-1010
Number analyzed (Participants) | 11026 | 11055
Participants | 45 | 40

12. Secondary Outcome: Number of Participants With Hospitalizations Associated With RT-PCR Confirmed Protocol-Defined ILI Caused by Any Seasonal Influenza A or B Virus Strains Regardless of Antigenic Match to Strains Selected for the Seasonal Vaccine
Description: as for outcome 5
Time Frame: 14 days post-vaccination through Day 181 (Month 6)
Population: as for outcome 6
Measure: Count of Participants; unit: Participants
Arm/Group | Fluarix Quadrivalent | mRNA-1010
Number analyzed (Participants) | 11026 | 11055
Participants | 3 | 3

13. Secondary Outcome: Geometric Mean Titer (GMT) of Anti-Hemagglutinin (HA) Antibodies at Day 29, as Measured by Hemagglutination Inhibition (HAI) Assay for Vaccine-matched Influenza A and B Strains
Description: Seasonal influenza A strains included H1N1 and H3N2 and seasonal influenza B strains included Victoria-lineage and Yamagata-lineage. 95% confidence interval (CI) was calculated based on the t-distribution of log-transformed values for GM titer, then back transformed to original scale for presentation.
Time Frame: Day 29
Population: PP Immunogenicity Set (PPIS) included all randomized participants in the biomarker subset who received any study intervention; had baseline and Day 29 antibody assessment via HAI assay; complied with the immunogenicity testing schedule, and had no major protocol deviations that impacted the immunogenicity assessment.
Measure: Geometric Mean (95% Confidence Interval); unit: titer
Arm/Group | Fluarix Quadrivalent | mRNA-1010
Number analyzed (Participants) | 408 | 444
titer
  Influenza A H1N1 Antibody | 105.34 [95.71 to 115.93] | 149.14 [135.47 to 164.19]
  Influenza A H3N2 Antibody | 85.99 [77.64 to 95.23] | 104.06 [94.35 to 114.77]
  Influenza B/ Yamagata Lineage | 140.50 [127.49 to 154.85] | 132.24 [121.25 to 144.23]
  Influenza B/ Victoria Lineage | 176.63 [162.42 to 192.08] | 139.91 [129.71 to 150.91]

14. Secondary Outcome: Percentage of Participants Reaching Seroconversion at Day 29, as Measured by HAI Assay for Vaccine-matched Influenza A and B Strains
Description: Seroconversion was defined as either a Baseline HAI titer <1:10 and a post-Baseline titer ≥1:40 or a Baseline HAI titer ≥1:10 and a minimum 4-fold rise in post-Baseline HAI antibody titer.
Time Frame: Day 29
Population: PPIS included all randomized participants in the biomarker subset who received any study intervention; had baseline and Day 29 antibody assessment via HAI assay; complied with the immunogenicity testing schedule, and had no major protocol deviations that impacted the immunogenicity assessment.
Measure: Number (95% Confidence Interval); unit: percentage of participants
Arm/Group | Fluarix Quadrivalent | mRNA-1010
Number analyzed (Participants) | 408 | 444
percentage of participants
  Influenza A H1N1 Antibody | 29.4 [25.03 to 34.09] | 44.8 [40.13 to 49.58]
  Influenza A H3N2 Antibody | 39.7 [34.93 to 44.64] | 52.0 [47.27 to 56.76]
  Influenza B/ Yamagata Lineage | 27.5 [23.18 to 32.06] | 26.6 [22.52 to 30.95]
  Influenza B/ Victoria Lineage | 22.8 [18.81 to 27.18] | 13.1 [10.07 to 16.56]

15. Secondary Outcome: Percentage of Participants With HAI Titer ≥ 1:40 at Day 29
Time Frame: Day 29
Population: as for outcome 14
Measure: Number (95% Confidence Interval); unit: percentage of participants
Arm/Group | Fluarix Quadrivalent | mRNA-1010
Number analyzed (Participants) | 408 | 444
percentage of participants
  Influenza A H1N1 Antibody | 90.0 [86.61 to 92.69] | 94.4 [91.80 to 96.32]
  Influenza A H3N2 Antibody | 85.5 [81.75 to 88.81] | 89.6 [86.42 to 92.31]
  Influenza B/ Yamagata Lineage | 94.6 [91.95 to 96.59] | 94.8 [92.33 to 96.69]
  Influenza B/ Victoria Lineage | 98.3 [96.50 to 99.31] | 98.0 [96.19 to 99.07]

16. Secondary Outcome: Geometric Mean Fold Rise (GMFR) of Anti-HA Antibodies at Day 29, as Measured by HAI Assay for Vaccine-matched Influenza A and B Strains
Description: The GMFR measures the changes in immunogenicity titers or levels from Baseline within participants. Seasonal influenza A included H1N1 and H3N2 and seasonal influenza B strains included Victoria-lineage and Yamagata-lineage. Fold-rise was calculated by dividing post-vaccination results by the baseline value. 95% CI for GMFR was calculated based on the t distribution of the differences in the log-transformed values between analysis timepoint and baseline, then back transformed to the original scale for presentation.
Time Frame: Baseline, Day 29
Population: as for outcome 14
Measure: Geometric Mean (95% Confidence Interval); unit: ratio
Arm/Group | Fluarix Quadrivalent | mRNA-1010
Number analyzed (Participants) | 408 | 444
ratio
  Influenza A H1N1 Antibody | 2.42 [2.22 to 2.64] | 3.42 [3.13 to 3.73]
  Influenza A H3N2 Antibody | 3.04 [2.79 to 3.30] | 3.74 [3.44 to 4.07]
  Influenza B/ Yamagata Lineage | 2.46 [2.26 to 2.69] | 2.28 [2.14 to 2.43]
  Influenza B/ Victoria Lineage | 2.07 [1.92 to 2.24] | 1.75 [1.65 to 1.85]

ADVERSE EVENTS:
Time Frame: Day 1 up to the end of the study (Day 361)
Description: The all-cause mortality was based on the randomization set. The serious and other (not including serious) adverse events were based on the safety set which consisted of all participants who received one dose of study vaccination. Participants were included in the vaccination group corresponding to the study intervention that they actually received.
Arm/Group | Fluarix Quadrivalent | mRNA-1010
All-Cause Mortality (participants affected / at risk) | 44/11250 | 45/11252
Serious Adverse Events (participants affected / at risk) | 495/11200 | 518/11210
Other Adverse Events (participants affected / at risk) | 603/11200 | 572/11210
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Fluarix Quadrivalent (N=11200) | mRNA-1010 (N=11210)
Abdominal abscess (Infections and infestations) | 0 (0) | 1 (1)
Abdominal sepsis (Infections and infestations) | 0 (0) | 1 (1)
Abscess limb (Infections and infestations) | 0 (0) | 1 (1)
Appendicitis (Infections and infestations) | 3 (3) | 5 (5)
Appendicitis perforated (Infections and infestations) | 2 (2) | 2 (2)
Arthritis bacterial (Infections and infestations) | 1 (1) | 1 (1)
Bacterial sepsis (Infections and infestations) | 1 (1) | 0 (0)
Bronchitis (Infections and infestations) | 3 (4) | 2 (2)
COVID-19 (Infections and infestations) | 8 (8) | 8 (8)
COVID-19 pneumonia (Infections and infestations) | 2 (2) | 2 (2)
Cellulitis (Infections and infestations) | 4 (4) | 9 (11)
Cellulitis staphylococcal (Infections and infestations) | 0 (0) | 2 (3)
Cholecystitis infective (Infections and infestations) | 0 (0) | 2 (2)
Clostridium difficile colitis (Infections and infestations) | 1 (1) | 0 (0)
Clostridium difficile infection (Infections and infestations) | 1 (1) | 0 (0)
Colonic abscess (Infections and infestations) | 1 (1) | 0 (0)
Complicated appendicitis (Infections and infestations) | 0 (0) | 2 (2)
Device related bacteraemia (Infections and infestations) | 1 (1) | 0 (0)
Device related infection (Infections and infestations) | 1 (1) | 1 (1)
Diverticulitis (Infections and infestations) | 7 (7) | 4 (5)
Endocarditis (Infections and infestations) | 1 (1) | 1 (1)
Epstein-Barr virus infection (Infections and infestations) | 1 (1) | 0 (0)
Escherichia infection (Infections and infestations) | 1 (1) | 0 (0)
Gangrene (Infections and infestations) | 1 (1) | 0 (0)
Gastroenteritis (Infections and infestations) | 2 (2) | 0 (0)
Gastroenteritis Escherichia coli (Infections and infestations) | 0 (0) | 1 (1)
Gastroenteritis viral (Infections and infestations) | 1 (1) | 0 (0)
Human anaplasmosis (Infections and infestations) | 1 (1) | 0 (0)
Influenza (Infections and infestations) | 2 (2) | 0 (0)
Intervertebral discitis (Infections and infestations) | 0 (0) | 1 (1)
Kidney infection (Infections and infestations) | 0 (0) | 2 (2)
Klebsiella infection (Infections and infestations) | 1 (1) | 0 (0)
Localised infection (Infections and infestations) | 1 (1) | 2 (2)
Meningitis (Infections and infestations) | 1 (1) | 0 (0)
Metapneumovirus infection (Infections and infestations) | 1 (1) | 1 (1)
Oral candidiasis (Infections and infestations) | 1 (1) | 0 (0)
Osteomyelitis (Infections and infestations) | 3 (3) | 4 (4)
Parainfluenzae viral bronchitis (Infections and infestations) | 0 (0) | 1 (1)
Periorbital cellulitis (Infections and infestations) | 1 (1) | 0 (0)
Perirectal abscess (Infections and infestations) | 0 (0) | 2 (2)
Peritonitis (Infections and infestations) | 1 (1) | 0 (0)
Pharyngitis streptococcal (Infections and infestations) | 2 (2) | 0 (0)
Pharyngolaryngeal abscess (Infections and infestations) | 0 (0) | 1 (1)
Pilonidal disease (Infections and infestations) | 1 (1) | 0 (0)
Pneumonia (Infections and infestations) | 21 (21) | 21 (22)
Pneumonia aspiration (Infections and infestations) | 1 (1) | 1 (1)
Pneumonia bacterial (Infections and infestations) | 2 (2) | 2 (2)
Pneumonia chlamydial (Infections and infestations) | 0 (0) | 1 (1)
Post procedural infection (Infections and infestations) | 1 (1) | 0 (0)
Post procedural sepsis (Infections and infestations) | 0 (0) | 1 (1)
Postoperative abscess (Infections and infestations) | 1 (1) | 1 (1)
Postoperative wound infection (Infections and infestations) | 1 (1) | 0 (0)
Prostatitis Escherichia coli (Infections and infestations) | 0 (0) | 1 (1)
Pyelonephritis (Infections and infestations) | 1 (1) | 0 (0)
Pyelonephritis acute (Infections and infestations) | 0 (0) | 2 (2)
Rectal abscess (Infections and infestations) | 0 (0) | 1 (1)
Respiratory syncytial virus infection (Infections and infestations) | 1 (1) | 0 (0)
Respiratory tract infection (Infections and infestations) | 0 (0) | 1 (1)
Rhinovirus infection (Infections and infestations) | 0 (0) | 3 (3)
Scrotal abscess (Infections and infestations) | 0 (0) | 1 (1)
Sepsis (Infections and infestations) | 9 (9) | 12 (12)
Septic shock (Infections and infestations) | 2 (2) | 1 (1)
Soft tissue infection (Infections and infestations) | 1 (1) | 0 (0)
Staphylococcal bacteraemia (Infections and infestations) | 0 (0) | 1 (1)
Staphylococcal skin infection (Infections and infestations) | 0 (0) | 2 (2)
Tularaemia (Infections and infestations) | 0 (0) | 1 (1)
Urinary tract infection (Infections and infestations) | 6 (6) | 11 (11)
Urosepsis (Infections and infestations) | 2 (2) | 2 (2)
Viral infection (Infections and infestations) | 1 (1) | 0 (0)
Vulval cellulitis (Infections and infestations) | 0 (0) | 1 (1)
Wound infection (Infections and infestations) | 0 (0) | 1 (1)
Acute leukaemia (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 (1) | 0 (0)
Adenocarcinoma gastric (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 (0) | 1 (1)
Adenocarcinoma of colon (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 (1) | 1 (1)
Adrenal adenoma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 (1) | 0 (0)
Basal cell carcinoma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 (0) | 1 (1)
Benign laryngeal neoplasm (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 (0) | 1 (1)
Benign neoplasm of testis (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 (1) | 0 (0)
Benign uterine neoplasm (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 (0) | 1 (1)
Bladder cancer (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 (0) | 2 (2)
Bladder transitional cell carcinoma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 (0) | 1 (1)
Bone cancer (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 (1) | 0 (0)
Bowen's disease (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 (0) | 1 (1)
Brain neoplasm malignant (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 (1) | 0 (0)
Breast cancer (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 8 (8) | 6 (6)
Breast cancer metastatic (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 (1) | 2 (2)
Breast cancer stage I (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 (0) | 1 (1)
Breast cancer stage II (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 (1) | 0 (0)
Carcinoid tumour pulmonary (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 (0) | 1 (1)
Chronic myeloid leukaemia (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 (0) | 1 (1)
Colon cancer (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 4 (4) | 3 (4)
Colon cancer stage III (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 (1) | 0 (0)
Colon cancer stage IV (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 (0) | 1 (1)
Cutaneous T-cell lymphoma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 (1) | 0 (0)
Endometrial adenocarcinoma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 (1) | 1 (1)
Endometrial cancer metastatic (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 (1) | 0 (0)
Epiglottic cancer (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 (1) | 0 (0)
Gallbladder cancer (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 (1) | 0 (0)
Gastric cancer (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 (0) | 1 (1)
Hepatic cancer (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 (1) | 0 (0)
Hepatocellular carcinoma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 (0) | 1 (1)
Intraductal proliferative breast lesion (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 (1) | 1 (1)
Invasive breast carcinoma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 (1) | 1 (1)
Invasive ductal breast carcinoma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 5 (5) | 1 (1)
Invasive lobular breast carcinoma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 (0) | 2 (2)
Laryngeal cancer (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 (1) | 0 (0)
Lentigo maligna (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 (0) | 1 (1)
Lobular breast carcinoma in situ (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 (0) | 1 (1)
Lung adenocarcinoma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 2 (2) | 0 (0)
Lung adenocarcinoma stage I (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 (0) | 1 (1)
Lung neoplasm malignant (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 (1) | 2 (2)
Malignant melanoma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 (1) | 0 (0)
Medullary thyroid cancer (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 (0) | 1 (1)
Metastases to central nervous system (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 (0) | 1 (1)
Metastases to liver (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 (0) | 1 (1)
Metastatic renal cell carcinoma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 (1) | 0 (0)
Non-small cell lung cancer (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 (0) | 1 (1)
Oesophageal carcinoma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 (1) | 1 (1)
Oesophageal squamous cell carcinoma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 (1) | 0 (0)
Oropharyngeal cancer (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 (0) | 1 (1)
Osteosarcoma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 (0) | 1 (1)
Ovarian adenoma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 (1) | 0 (0)
Ovarian cancer metastatic (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 (0) | 1 (1)
Pancreatic carcinoma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 (0) | 1 (1)
Pancreatic carcinoma metastatic (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 (0) | 1 (1)
Plasma cell myeloma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 (0) | 1 (1)
Primary myelofibrosis (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 (1) | 0 (0)
Prostate cancer (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 12 (12) | 4 (4)
Prostate cancer metastatic (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 (1) | 1 (1)
Rectal adenocarcinoma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 (0) | 1 (1)
Rectal cancer (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 (1) | 0 (0)
Renal cell carcinoma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 2 (2) | 1 (1)
Small cell carcinoma of the cervix (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 (1) | 0 (0)
Small intestine adenocarcinoma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 (1) | 0 (0)
Small intestine neuroendocrine tumour (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 (0) | 1 (1)
Squamous cell carcinoma of lung (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 (1) | 0 (0)
Transitional cell carcinoma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 (0) | 2 (2)
Uterine leiomyoma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 (1) | 1 (1)
Vulval cancer stage 0 (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 (0) | 1 (1)
Anaemia (Blood and lymphatic system disorders) | 1 (1) | 3 (3)
Blood loss anaemia (Blood and lymphatic system disorders) | 1 (1) | 2 (2)
Hypochromic anaemia (Blood and lymphatic system disorders) | 0 (0) | 1 (1)
Immune thrombocytopenia (Blood and lymphatic system disorders) | 0 (0) | 2 (2)
Iron deficiency anaemia (Blood and lymphatic system disorders) | 0 (0) | 1 (1)
Leukocytosis (Blood and lymphatic system disorders) | 1 (1) | 1 (1)
Methaemoglobinaemia (Blood and lymphatic system disorders) | 0 (0) | 1 (1)
Thrombocytosis (Blood and lymphatic system disorders) | 1 (1) | 0 (0)
Anaphylactic reaction (Immune system disorders) | 3 (3) | 0 (0)
Drug hypersensitivity (Immune system disorders) | 0 (0) | 1 (1)
Goitre (Endocrine disorders) | 1 (1) | 0 (0)
Hyperparathyroidism (Endocrine disorders) | 0 (0) | 1 (1)
Hyperthyroidism (Endocrine disorders) | 0 (0) | 1 (1)
Inappropriate antidiuretic hormone secretion (Endocrine disorders) | 0 (0) | 1 (1)
Primary hyperaldosteronism (Endocrine disorders) | 0 (0) | 1 (1)
Alcoholic ketoacidosis (Metabolism and nutrition disorders) | 0 (0) | 1 (1)
Dehydration (Metabolism and nutrition disorders) | 3 (3) | 0 (0)
Diabetic complication (Metabolism and nutrition disorders) | 0 (0) | 2 (2)
Diabetic ketoacidosis (Metabolism and nutrition disorders) | 2 (5) | 1 (1)
Fluid retention (Metabolism and nutrition disorders) | 1 (1) | 0 (0)
Hypercalcaemia (Metabolism and nutrition disorders) | 1 (1) | 1 (1)
Hyperglycaemia (Metabolism and nutrition disorders) | 1 (1) | 0 (0)
Hyperglycaemic hyperosmolar nonketotic syndrome (Metabolism and nutrition disorders) | 2 (3) | 1 (1)
Hyperkalaemia (Metabolism and nutrition disorders) | 1 (1) | 0 (0)
Hypervolaemia (Metabolism and nutrition disorders) | 1 (1) | 0 (0)
Hypocalcaemia (Metabolism and nutrition disorders) | 0 (0) | 1 (1)
Hypoglycaemia (Metabolism and nutrition disorders) | 1 (1) | 0 (0)
Hypokalaemia (Metabolism and nutrition disorders) | 2 (2) | 1 (1)
Hypomagnesaemia (Metabolism and nutrition disorders) | 1 (1) | 0 (0)
Hyponatraemia (Metabolism and nutrition disorders) | 2 (2) | 4 (4)
Hypovolaemia (Metabolism and nutrition disorders) | 1 (1) | 0 (0)
Lactic acidosis (Metabolism and nutrition disorders) | 1 (1) | 0 (0)
Malnutrition (Metabolism and nutrition disorders) | 1 (1) | 0 (0)
Obesity (Metabolism and nutrition disorders) | 3 (3) | 2 (2)
Steroid diabetes (Metabolism and nutrition disorders) | 1 (1) | 0 (0)
Type 2 diabetes mellitus (Metabolism and nutrition disorders) | 2 (4) | 2 (2)
Acute psychosis (Psychiatric disorders) | 1 (1) | 0 (0)
Affective disorder (Psychiatric disorders) | 1 (1) | 0 (0)
Alcohol abuse (Psychiatric disorders) | 1 (1) | 0 (0)
Alcohol use disorder (Psychiatric disorders) | 1 (1) | 1 (1)
Alcohol withdrawal syndrome (Psychiatric disorders) | 0 (0) | 1 (1)
Anxiety (Psychiatric disorders) | 2 (2) | 0 (0)
Bipolar disorder (Psychiatric disorders) | 1 (1) | 0 (0)
Completed suicide (Psychiatric disorders) | 0 (0) | 1 (1)
Confusional state (Psychiatric disorders) | 1 (1) | 0 (0)
Delirium (Psychiatric disorders) | 0 (0) | 1 (1)
Depression (Psychiatric disorders) | 1 (1) | 2 (2)
Depression suicidal (Psychiatric disorders) | 1 (1) | 1 (1)
Drug dependence (Psychiatric disorders) | 1 (1) | 1 (1)
Major depression (Psychiatric disorders) | 0 (0) | 1 (1)
Mental status changes (Psychiatric disorders) | 0 (0) | 1 (1)
Mixed anxiety and depressive disorder (Psychiatric disorders) | 1 (1) | 0 (0)
Post-traumatic stress disorder (Psychiatric disorders) | 1 (1) | 0 (0)
Psychotic disorder (Psychiatric disorders) | 1 (1) | 0 (0)
Schizoaffective disorder (Psychiatric disorders) | 0 (0) | 1 (1)
Substance abuse (Psychiatric disorders) | 3 (3) | 0 (0)
Suicidal ideation (Psychiatric disorders) | 0 (0) | 1 (1)
Amyotrophic lateral sclerosis (Nervous system disorders) | 0 (0) | 1 (1)
Carotid artery disease (Nervous system disorders) | 0 (0) | 1 (1)
Carotid artery occlusion (Nervous system disorders) | 0 (0) | 1 (1)
Carotid artery stenosis (Nervous system disorders) | 1 (1) | 1 (1)
Cerebellar infarction (Nervous system disorders) | 1 (1) | 0 (0)
Cerebellar stroke (Nervous system disorders) | 0 (0) | 1 (1)
Cerebral artery embolism (Nervous system disorders) | 1 (1) | 0 (0)
Cerebral infarction (Nervous system disorders) | 1 (1) | 1 (1)
Cerebral venous sinus thrombosis (Nervous system disorders) | 1 (1) | 0 (0)
Cerebral ventricle dilatation (Nervous system disorders) | 0 (0) | 1 (1)
Cerebrospinal fluid leakage (Nervous system disorders) | 0 (0) | 1 (1)
Cerebrovascular accident (Nervous system disorders) | 14 (14) | 16 (16)
Cervical radiculopathy (Nervous system disorders) | 1 (1) | 0 (0)
Cranial nerve paralysis (Nervous system disorders) | 0 (0) | 1 (1)
Dementia (Nervous system disorders) | 2 (2) | 0 (0)
Dementia Alzheimer's type (Nervous system disorders) | 1 (1) | 0 (0)
Dizziness (Nervous system disorders) | 4 (4) | 1 (1)
Embolic stroke (Nervous system disorders) | 1 (1) | 0 (0)
Encephalopathy (Nervous system disorders) | 2 (3) | 0 (0)
Generalised tonic-clonic seizure (Nervous system disorders) | 0 (0) | 1 (1)
Haemorrhagic stroke (Nervous system disorders) | 0 (0) | 1 (1)
Hemiparesis (Nervous system disorders) | 0 (0) | 1 (1)
Hypoaesthesia (Nervous system disorders) | 1 (1) | 0 (0)
Ischaemic stroke (Nervous system disorders) | 5 (5) | 2 (2)
Lacunar infarction (Nervous system disorders) | 0 (0) | 1 (1)
Lacunar stroke (Nervous system disorders) | 2 (2) | 0 (0)
Lumbar radiculopathy (Nervous system disorders) | 1 (1) | 1 (1)
Metabolic encephalopathy (Nervous system disorders) | 2 (2) | 1 (1)
Migraine with aura (Nervous system disorders) | 0 (0) | 1 (1)
Multiple sclerosis (Nervous system disorders) | 1 (1) | 0 (0)
Multiple sclerosis relapse (Nervous system disorders) | 1 (1) | 0 (0)
Myelopathy (Nervous system disorders) | 2 (2) | 0 (0)
Nerve compression (Nervous system disorders) | 1 (1) | 1 (1)
Paraesthesia (Nervous system disorders) | 0 (0) | 1 (1)
Piriformis syndrome (Nervous system disorders) | 1 (1) | 0 (0)
Post herpetic neuralgia (Nervous system disorders) | 1 (1) | 0 (0)
Presyncope (Nervous system disorders) | 1 (1) | 0 (0)
Radial nerve palsy (Nervous system disorders) | 0 (0) | 1 (1)
Sciatica (Nervous system disorders) | 1 (1) | 0 (0)
Seizure (Nervous system disorders) | 2 (2) | 3 (3)
Spinal cord disorder (Nervous system disorders) | 1 (1) | 0 (0)
Spinal cord haematoma (Nervous system disorders) | 0 (0) | 1 (1)
Spinal meningeal cyst (Nervous system disorders) | 0 (0) | 1 (1)
Status epilepticus (Nervous system disorders) | 0 (0) | 1 (1)
Subarachnoid haemorrhage (Nervous system disorders) | 0 (0) | 1 (1)
Syncope (Nervous system disorders) | 6 (7) | 5 (5)
Transient global amnesia (Nervous system disorders) | 0 (0) | 1 (1)
Transient ischaemic attack (Nervous system disorders) | 6 (6) | 2 (2)
Tremor (Nervous system disorders) | 0 (0) | 1 (1)
Vertebrobasilar stroke (Nervous system disorders) | 1 (1) | 0 (0)
Disorder of orbit (Eye disorders) | 1 (1) | 0 (0)
Retinal artery occlusion (Eye disorders) | 0 (0) | 1 (1)
Vision blurred (Eye disorders) | 0 (0) | 1 (1)
Vitreous haemorrhage (Eye disorders) | 0 (0) | 1 (1)
Vertigo (Ear and labyrinth disorders) | 5 (5) | 0 (0)
Vertigo positional (Ear and labyrinth disorders) | 0 (0) | 1 (1)
Acute left ventricular failure (Cardiac disorders) | 2 (2) | 2 (2)
Acute myocardial infarction (Cardiac disorders) | 11 (12) | 12 (12)
Angina pectoris (Cardiac disorders) | 5 (5) | 3 (3)
Angina unstable (Cardiac disorders) | 3 (3) | 2 (3)
Aortic valve incompetence (Cardiac disorders) | 0 (0) | 1 (1)
Aortic valve stenosis (Cardiac disorders) | 1 (1) | 0 (0)
Arrhythmia (Cardiac disorders) | 1 (1) | 0 (0)
Arteriosclerosis coronary artery (Cardiac disorders) | 0 (0) | 1 (1)
Atrial fibrillation (Cardiac disorders) | 14 (15) | 16 (19)
Atrial flutter (Cardiac disorders) | 1 (1) | 1 (1)
Atrioventricular block (Cardiac disorders) | 1 (1) | 0 (0)
Bradycardia (Cardiac disorders) | 0 (0) | 3 (3)
Cardiac arrest (Cardiac disorders) | 3 (3) | 3 (3)
Cardiac disorder (Cardiac disorders) | 0 (0) | 1 (1)
Cardiac failure (Cardiac disorders) | 5 (5) | 2 (2)
Cardiac failure acute (Cardiac disorders) | 5 (5) | 2 (3)
Cardiac failure chronic (Cardiac disorders) | 0 (0) | 1 (1)
Cardiac failure congestive (Cardiac disorders) | 10 (11) | 11 (14)
Cardio-respiratory arrest (Cardiac disorders) | 3 (3) | 0 (0)
Cardiogenic shock (Cardiac disorders) | 0 (0) | 1 (1)
Cardiomyopathy (Cardiac disorders) | 0 (0) | 1 (1)
Cardiopulmonary failure (Cardiac disorders) | 0 (0) | 1 (1)
Coronary artery aneurysm (Cardiac disorders) | 0 (0) | 1 (1)
Coronary artery disease (Cardiac disorders) | 9 (9) | 8 (8)
Coronary artery dissection (Cardiac disorders) | 1 (1) | 0 (0)
Coronary artery occlusion (Cardiac disorders) | 1 (1) | 0 (0)
Coronary artery stenosis (Cardiac disorders) | 1 (1) | 1 (1)
Intracardiac thrombus (Cardiac disorders) | 1 (1) | 0 (0)
Left ventricular failure (Cardiac disorders) | 1 (1) | 0 (0)
Mitral valve incompetence (Cardiac disorders) | 2 (2) | 1 (1)
Mitral valve prolapse (Cardiac disorders) | 0 (0) | 2 (2)
Myocardial infarction (Cardiac disorders) | 9 (9) | 12 (12)
Myocardial ischaemia (Cardiac disorders) | 1 (1) | 0 (0)
Myocarditis (Cardiac disorders) | 1 (1) | 0 (0)
Myopericarditis (Cardiac disorders) | 1 (1) | 0 (0)
Pericardial effusion (Cardiac disorders) | 1 (1) | 0 (0)
Pericarditis (Cardiac disorders) | 1 (1) | 4 (4)
Sinus arrhythmia (Cardiac disorders) | 1 (1) | 0 (0)
Sinus node dysfunction (Cardiac disorders) | 3 (3) | 0 (0)
Supraventricular tachycardia (Cardiac disorders) | 2 (2) | 2 (2)
Tachycardia (Cardiac disorders) | 0 (0) | 3 (3)
Ventricular arrhythmia (Cardiac disorders) | 0 (0) | 1 (1)
Ventricular tachycardia (Cardiac disorders) | 0 (0) | 2 (2)
Aortic aneurysm (Vascular disorders) | 4 (4) | 1 (1)
Aortic dissection (Vascular disorders) | 1 (1) | 1 (1)
Aortic stenosis (Vascular disorders) | 1 (1) | 2 (2)
Arteriosclerosis (Vascular disorders) | 0 (0) | 1 (1)
Deep vein thrombosis (Vascular disorders) | 5 (5) | 4 (4)
Dry gangrene (Vascular disorders) | 0 (0) | 1 (1)
Embolism (Vascular disorders) | 1 (1) | 0 (0)
Giant cell arteritis (Vascular disorders) | 1 (1) | 0 (0)
Hypertension (Vascular disorders) | 4 (4) | 5 (5)
Hypertensive crisis (Vascular disorders) | 2 (2) | 2 (2)
Hypertensive emergency (Vascular disorders) | 1 (2) | 0 (0)
Hypertensive urgency (Vascular disorders) | 3 (3) | 1 (1)
Hypotension (Vascular disorders) | 4 (4) | 1 (1)
Peripheral arterial occlusive disease (Vascular disorders) | 3 (4) | 4 (4)
Peripheral artery occlusion (Vascular disorders) | 0 (0) | 1 (1)
Peripheral artery stenosis (Vascular disorders) | 0 (0) | 2 (2)
Peripheral artery thrombosis (Vascular disorders) | 0 (0) | 1 (1)
Peripheral ischaemia (Vascular disorders) | 0 (0) | 1 (1)
Peripheral vascular disorder (Vascular disorders) | 0 (0) | 2 (2)
Shock (Vascular disorders) | 1 (1) | 0 (0)
Vascular stenosis (Vascular disorders) | 0 (0) | 1 (1)
Acute pulmonary oedema (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 1 (1)
Acute respiratory distress syndrome (Respiratory, thoracic and mediastinal disorders) | 1 (1) | 0 (0)
Acute respiratory failure (Respiratory, thoracic and mediastinal disorders) | 10 (11) | 8 (11)
Asthma (Respiratory, thoracic and mediastinal disorders) | 2 (2) | 2 (2)
Bronchiectasis (Respiratory, thoracic and mediastinal disorders) | 1 (1) | 1 (1)
Chronic obstructive pulmonary disease (Respiratory, thoracic and mediastinal disorders) | 14 (14) | 19 (25)
Cough (Respiratory, thoracic and mediastinal disorders) | 2 (2) | 0 (0)
Dyspnoea (Respiratory, thoracic and mediastinal disorders) | 4 (4) | 1 (1)
Emphysema (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 1 (2)
Haemothorax (Respiratory, thoracic and mediastinal disorders) | 1 (1) | 1 (1)
Hypercapnia (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 1 (1)
Hypoxia (Respiratory, thoracic and mediastinal disorders) | 1 (1) | 0 (0)
Interstitial lung disease (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 1 (1)
Nasal septum deviation (Respiratory, thoracic and mediastinal disorders) | 1 (1) | 0 (0)
Organising pneumonia (Respiratory, thoracic and mediastinal disorders) | 1 (1) | 0 (0)
Pleural effusion (Respiratory, thoracic and mediastinal disorders) | 2 (2) | 1 (1)
Pneumothorax (Respiratory, thoracic and mediastinal disorders) | 1 (1) | 3 (3)
Pneumothorax spontaneous (Respiratory, thoracic and mediastinal disorders) | 1 (1) | 0 (0)
Productive cough (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 1 (1)
Pulmonary embolism (Respiratory, thoracic and mediastinal disorders) | 12 (12) | 8 (8)
Pulmonary fibrosis (Respiratory, thoracic and mediastinal disorders) | 1 (1) | 0 (0)
Pulmonary hypertension (Respiratory, thoracic and mediastinal disorders) | 1 (1) | 2 (2)
Pulmonary mass (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 1 (1)
Pulmonary oedema (Respiratory, thoracic and mediastinal disorders) | 1 (1) | 0 (0)
Respiratory failure (Respiratory, thoracic and mediastinal disorders) | 1 (1) | 3 (3)
Sleep apnoea syndrome (Respiratory, thoracic and mediastinal disorders) | 1 (1) | 0 (0)
Abdominal adhesions (Gastrointestinal disorders) | 1 (1) | 0 (0)
Abdominal discomfort (Gastrointestinal disorders) | 1 (1) | 0 (0)
Abdominal hernia (Gastrointestinal disorders) | 1 (1) | 0 (0)
Abdominal pain (Gastrointestinal disorders) | 0 (0) | 5 (6)
Ascites (Gastrointestinal disorders) | 1 (1) | 0 (0)
Colitis (Gastrointestinal disorders) | 3 (3) | 5 (5)
Colitis ischaemic (Gastrointestinal disorders) | 0 (0) | 1 (1)
Colitis ulcerative (Gastrointestinal disorders) | 0 (0) | 1 (1)
Constipation (Gastrointestinal disorders) | 2 (2) | 0 (0)
Diarrhoea (Gastrointestinal disorders) | 1 (1) | 0 (0)
Diverticular perforation (Gastrointestinal disorders) | 1 (1) | 0 (0)
Diverticulum intestinal (Gastrointestinal disorders) | 1 (1) | 0 (0)
Duodenal ulcer perforation (Gastrointestinal disorders) | 1 (1) | 0 (0)
Duodenitis (Gastrointestinal disorders) | 0 (0) | 1 (1)
Enteritis (Gastrointestinal disorders) | 0 (0) | 1 (1)
Gastric ulcer (Gastrointestinal disorders) | 1 (1) | 2 (2)
Gastritis (Gastrointestinal disorders) | 1 (1) | 1 (1)
Gastritis alcoholic (Gastrointestinal disorders) | 0 (0) | 1 (1)
Gastrointestinal disorder (Gastrointestinal disorders) | 1 (1) | 0 (0)
Gastrointestinal haemorrhage (Gastrointestinal disorders) | 1 (1) | 0 (0)
Gastrooesophageal reflux disease (Gastrointestinal disorders) | 2 (2) | 1 (1)
Hiatus hernia (Gastrointestinal disorders) | 0 (0) | 3 (3)
Ileus (Gastrointestinal disorders) | 2 (2) | 1 (1)
Impaired gastric emptying (Gastrointestinal disorders) | 1 (1) | 0 (0)
Incarcerated inguinal hernia (Gastrointestinal disorders) | 0 (0) | 1 (1)
Inguinal hernia (Gastrointestinal disorders) | 1 (1) | 0 (0)
Intestinal ischaemia (Gastrointestinal disorders) | 0 (0) | 1 (1)
Intestinal mass (Gastrointestinal disorders) | 1 (1) | 0 (0)
Intestinal obstruction (Gastrointestinal disorders) | 1 (1) | 4 (4)
Intestinal perforation (Gastrointestinal disorders) | 2 (2) | 1 (1)
Intussusception (Gastrointestinal disorders) | 0 (0) | 2 (2)
Large intestine perforation (Gastrointestinal disorders) | 0 (0) | 1 (1)
Large intestine polyp (Gastrointestinal disorders) | 1 (1) | 0 (0)
Lower gastrointestinal haemorrhage (Gastrointestinal disorders) | 0 (0) | 1 (1)
Melaena (Gastrointestinal disorders) | 1 (1) | 0 (0)
Nausea (Gastrointestinal disorders) | 2 (2) | 1 (1)
Oesophagitis (Gastrointestinal disorders) | 0 (0) | 1 (1)
Pancreatitis (Gastrointestinal disorders) | 1 (1) | 3 (3)
Pancreatitis acute (Gastrointestinal disorders) | 3 (3) | 2 (2)
Pancreatitis chronic (Gastrointestinal disorders) | 1 (1) | 1 (1)
Rectal haemorrhage (Gastrointestinal disorders) | 0 (0) | 1 (1)
Small intestinal obstruction (Gastrointestinal disorders) | 3 (3) | 7 (7)
Small intestinal perforation (Gastrointestinal disorders) | 1 (1) | 2 (2)
Umbilical hernia (Gastrointestinal disorders) | 2 (2) | 0 (0)
Umbilical hernia perforation (Gastrointestinal disorders) | 0 (0) | 1 (1)
Upper gastrointestinal haemorrhage (Gastrointestinal disorders) | 1 (1) | 2 (2)
Volvulus (Gastrointestinal disorders) | 0 (0) | 1 (1)
Vomiting (Gastrointestinal disorders) | 0 (0) | 2 (2)
Bile duct stone (Hepatobiliary disorders) | 1 (1) | 1 (1)
Biliary colic (Hepatobiliary disorders) | 1 (1) | 1 (1)
Cholangitis (Hepatobiliary disorders) | 1 (1) | 0 (0)
Cholecystitis (Hepatobiliary disorders) | 2 (2) | 1 (1)
Cholecystitis acute (Hepatobiliary disorders) | 3 (3) | 3 (3)
Cholelithiasis (Hepatobiliary disorders) | 5 (5) | 4 (4)
Hepatic failure (Hepatobiliary disorders) | 1 (1) | 0 (0)
Hepatorenal failure (Hepatobiliary disorders) | 1 (1) | 0 (0)
Angioedema (Skin and subcutaneous tissue disorders) | 1 (1) | 1 (1)
Dermatitis allergic (Skin and subcutaneous tissue disorders) | 0 (0) | 1 (1)
Excessive skin (Skin and subcutaneous tissue disorders) | 0 (0) | 1 (1)
Skin lesion (Skin and subcutaneous tissue disorders) | 1 (1) | 0 (0)
Arthralgia (Musculoskeletal and connective tissue disorders) | 1 (1) | 1 (1)
Arthritis (Musculoskeletal and connective tissue disorders) | 0 (0) | 3 (3)
Arthropathy (Musculoskeletal and connective tissue disorders) | 0 (0) | 1 (1)
Back pain (Musculoskeletal and connective tissue disorders) | 2 (2) | 3 (3)
Bone demineralisation (Musculoskeletal and connective tissue disorders) | 0 (0) | 1 (1)
Cervical spinal stenosis (Musculoskeletal and connective tissue disorders) | 2 (2) | 1 (1)
Exostosis (Musculoskeletal and connective tissue disorders) | 1 (1) | 0 (0)
Foot deformity (Musculoskeletal and connective tissue disorders) | 1 (1) | 1 (1)
Fracture nonunion (Musculoskeletal and connective tissue disorders) | 1 (1) | 0 (0)
Intervertebral disc degeneration (Musculoskeletal and connective tissue disorders) | 3 (3) | 2 (2)
Intervertebral disc disorder (Musculoskeletal and connective tissue disorders) | 1 (1) | 2 (2)
Intervertebral disc protrusion (Musculoskeletal and connective tissue disorders) | 2 (2) | 2 (2)
Lumbar spinal stenosis (Musculoskeletal and connective tissue disorders) | 1 (1) | 2 (2)
Muscle spasms (Musculoskeletal and connective tissue disorders) | 1 (1) | 0 (0)
Muscular weakness (Musculoskeletal and connective tissue disorders) | 0 (0) | 1 (1)
Musculoskeletal chest pain (Musculoskeletal and connective tissue disorders) | 1 (1) | 2 (2)
Neck pain (Musculoskeletal and connective tissue disorders) | 1 (1) | 0 (0)
Osteoarthritis (Musculoskeletal and connective tissue disorders) | 22 (22) | 12 (12)
Osteochondrosis (Musculoskeletal and connective tissue disorders) | 0 (0) | 1 (1)
Polyarthritis (Musculoskeletal and connective tissue disorders) | 0 (0) | 1 (1)
Polymyositis (Musculoskeletal and connective tissue disorders) | 0 (0) | 1 (1)
Rhabdomyolysis (Musculoskeletal and connective tissue disorders) | 1 (1) | 1 (1)
Rotator cuff syndrome (Musculoskeletal and connective tissue disorders) | 1 (1) | 1 (1)
Soft tissue necrosis (Musculoskeletal and connective tissue disorders) | 0 (0) | 1 (1)
Spinal osteoarthritis (Musculoskeletal and connective tissue disorders) | 4 (4) | 0 (0)
Spinal stenosis (Musculoskeletal and connective tissue disorders) | 3 (3) | 2 (2)
Spondylolisthesis (Musculoskeletal and connective tissue disorders) | 1 (1) | 0 (0)
Vertebral foraminal stenosis (Musculoskeletal and connective tissue disorders) | 0 (0) | 1 (1)
Acute kidney injury (Renal and urinary disorders) | 14 (15) | 12 (12)
Bladder stenosis (Renal and urinary disorders) | 1 (1) | 0 (0)
Calculus urinary (Renal and urinary disorders) | 0 (0) | 1 (1)
Chronic kidney disease (Renal and urinary disorders) | 2 (2) | 0 (0)
Hydronephrosis (Renal and urinary disorders) | 1 (1) | 1 (1)
Nephrolithiasis (Renal and urinary disorders) | 2 (2) | 5 (6)
Renal cyst (Renal and urinary disorders) | 1 (1) | 0 (0)
Renal failure (Renal and urinary disorders) | 1 (1) | 3 (3)
Renal impairment (Renal and urinary disorders) | 1 (1) | 1 (1)
Stress urinary incontinence (Renal and urinary disorders) | 1 (1) | 0 (0)
Ureterolithiasis (Renal and urinary disorders) | 1 (1) | 0 (0)
Urinary retention (Renal and urinary disorders) | 1 (1) | 0 (0)
Benign prostatic hyperplasia (Reproductive system and breast disorders) | 1 (1) | 1 (1)
Prostatomegaly (Reproductive system and breast disorders) | 0 (0) | 1 (1)
Vaginal haemorrhage (Reproductive system and breast disorders) | 0 (0) | 1 (1)
Congenital cystic kidney disease (Congenital, familial and genetic disorders) | 0 (0) | 1 (1)
Asthenia (General disorders) | 1 (1) | 1 (1)
Chest discomfort (General disorders) | 0 (0) | 1 (1)
Chest pain (General disorders) | 4 (4) | 2 (2)
Death (General disorders) | 4 (4) | 8 (8)
Drug withdrawal syndrome (General disorders) | 0 (0) | 1 (1)
Generalised oedema (General disorders) | 0 (0) | 1 (1)
Non-cardiac chest pain (General disorders) | 4 (4) | 5 (5)
Oedema peripheral (General disorders) | 0 (0) | 1 (1)
Pain (General disorders) | 1 (1) | 1 (1)
Pyrexia (General disorders) | 2 (2) | 1 (1)
Stent-graft endoleak (General disorders) | 0 (0) | 1 (1)
Strangulated hernia (General disorders) | 1 (1) | 0 (0)
Sudden death (General disorders) | 1 (1) | 3 (3)
Blood potassium decreased (Investigations) | 1 (1) | 0 (0)
Hepatic enzyme abnormal (Investigations) | 0 (0) | 1 (1)
Hepatic enzyme increased (Investigations) | 1 (1) | 0 (0)
International normalised ratio abnormal (Investigations) | 0 (0) | 1 (1)
Liver function test abnormal (Investigations) | 0 (0) | 1 (1)
Prostatic specific antigen increased (Investigations) | 0 (0) | 1 (1)
Troponin increased (Investigations) | 1 (1) | 0 (0)
Weight increased (Investigations) | 0 (0) | 1 (1)
White blood cell count increased (Investigations) | 1 (1) | 0 (0)
Accidental overdose (Injury, poisoning and procedural complications) | 1 (1) | 2 (3)
Acetabulum fracture (Injury, poisoning and procedural complications) | 1 (1) | 0 (0)
Alcohol poisoning (Injury, poisoning and procedural complications) | 1 (1) | 0 (0)
Anastomotic ulcer (Injury, poisoning and procedural complications) | 1 (1) | 0 (0)
Animal bite (Injury, poisoning and procedural complications) | 1 (1) | 0 (0)
Ankle fracture (Injury, poisoning and procedural complications) | 3 (3) | 4 (4)
Bronchitis chemical (Injury, poisoning and procedural complications) | 0 (0) | 1 (1)
Cervical vertebral fracture (Injury, poisoning and procedural complications) | 2 (2) | 0 (0)
Concussion (Injury, poisoning and procedural complications) | 2 (2) | 0 (0)
Contusion (Injury, poisoning and procedural complications) | 1 (1) | 0 (0)
Craniocerebral injury (Injury, poisoning and procedural complications) | 0 (0) | 1 (1)
Facial bones fracture (Injury, poisoning and procedural complications) | 0 (0) | 1 (1)
Fall (Injury, poisoning and procedural complications) | 1 (1) | 2 (2)
Femoral neck fracture (Injury, poisoning and procedural complications) | 0 (0) | 1 (1)
Femoral nerve injury (Injury, poisoning and procedural complications) | 1 (1) | 0 (0)
Femur fracture (Injury, poisoning and procedural complications) | 1 (1) | 4 (4)
Fibula fracture (Injury, poisoning and procedural complications) | 1 (1) | 1 (1)
Foot fracture (Injury, poisoning and procedural complications) | 2 (2) | 0 (0)
Forearm fracture (Injury, poisoning and procedural complications) | 1 (1) | 1 (1)
Fracture displacement (Injury, poisoning and procedural complications) | 1 (1) | 1 (1)
Gastrointestinal procedural complication (Injury, poisoning and procedural complications) | 0 (0) | 1 (1)
Gun shot wound (Injury, poisoning and procedural complications) | 2 (2) | 0 (0)
Hand fracture (Injury, poisoning and procedural complications) | 0 (0) | 1 (1)
Head injury (Injury, poisoning and procedural complications) | 1 (1) | 0 (0)
Heat exhaustion (Injury, poisoning and procedural complications) | 1 (1) | 0 (0)
Hip fracture (Injury, poisoning and procedural complications) | 1 (1) | 4 (4)
Humerus fracture (Injury, poisoning and procedural complications) | 0 (0) | 2 (2)
Injury (Injury, poisoning and procedural complications) | 1 (1) | 0 (0)
Joint dislocation (Injury, poisoning and procedural complications) | 0 (0) | 2 (3)
Limb crushing injury (Injury, poisoning and procedural complications) | 1 (1) | 0 (0)
Limb injury (Injury, poisoning and procedural complications) | 1 (1) | 0 (0)
Lumbar vertebral fracture (Injury, poisoning and procedural complications) | 2 (2) | 1 (1)
Multiple injuries (Injury, poisoning and procedural complications) | 1 (1) | 0 (0)
Overdose (Injury, poisoning and procedural complications) | 0 (0) | 2 (2)
Patella fracture (Injury, poisoning and procedural complications) | 1 (1) | 0 (0)
Pelvic fracture (Injury, poisoning and procedural complications) | 0 (0) | 1 (1)
Periprosthetic fracture (Injury, poisoning and procedural complications) | 1 (1) | 2 (2)
Post procedural complication (Injury, poisoning and procedural complications) | 2 (2) | 1 (1)
Post procedural haemorrhage (Injury, poisoning and procedural complications) | 1 (1) | 1 (1)
Procedural pain (Injury, poisoning and procedural complications) | 1 (1) | 3 (3)
Rib fracture (Injury, poisoning and procedural complications) | 5 (5) | 3 (3)
Road traffic accident (Injury, poisoning and procedural complications) | 4 (4) | 2 (2)
Sacroiliac fracture (Injury, poisoning and procedural complications) | 0 (0) | 1 (1)
Skin abrasion (Injury, poisoning and procedural complications) | 1 (1) | 0 (0)
Skin laceration (Injury, poisoning and procedural complications) | 2 (2) | 0 (0)
Skull fracture (Injury, poisoning and procedural complications) | 0 (0) | 1 (1)
Snake bite (Injury, poisoning and procedural complications) | 1 (1) | 0 (0)
Spinal compression fracture (Injury, poisoning and procedural complications) | 1 (1) | 1 (1)
Spinal cord injury (Injury, poisoning and procedural complications) | 0 (0) | 1 (1)
Spinal fracture (Injury, poisoning and procedural complications) | 1 (1) | 0 (0)
Splenic rupture (Injury, poisoning and procedural complications) | 1 (1) | 1 (1)
Subdural haematoma (Injury, poisoning and procedural complications) | 1 (1) | 1 (1)
Tendon rupture (Injury, poisoning and procedural complications) | 1 (1) | 0 (0)
Thoracic vertebral fracture (Injury, poisoning and procedural complications) | 1 (1) | 1 (1)
Tibia fracture (Injury, poisoning and procedural complications) | 2 (2) | 0 (0)
Toxicity to various agents (Injury, poisoning and procedural complications) | 0 (0) | 1 (1)
Transplant failure (Injury, poisoning and procedural complications) | 1 (1) | 0 (0)
Traumatic haemothorax (Injury, poisoning and procedural complications) | 1 (1) | 0 (0)
Traumatic liver injury (Injury, poisoning and procedural complications) | 1 (1) | 1 (1)
Traumatic lung injury (Injury, poisoning and procedural complications) | 1 (1) | 0 (0)
Ulna fracture (Injury, poisoning and procedural complications) | 1 (1) | 0 (0)
Upper limb fracture (Injury, poisoning and procedural complications) | 1 (1) | 2 (2)
Vascular graft complication (Injury, poisoning and procedural complications) | 0 (0) | 1 (3)
Wrist fracture (Injury, poisoning and procedural complications) | 1 (1) | 0 (0)
OTHER ADVERSE EVENTS (reported when occurring in more than 5% of participants in an arm); cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Fluarix Quadrivalent (N=11200) | mRNA-1010 (N=11210)
COVID-19 (Infections and infestations) | 603 (621) | 572 (581)

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes

DOCUMENTS (2):
  • Study Protocol (2023-02-02): https://cdn.clinicaltrials.gov/large-docs/39/NCT05566639/Prot_000.pdf
  • Statistical Analysis Plan (2023-02-23): https://cdn.clinicaltrials.gov/large-docs/39/NCT05566639/SAP_001.pdf